CLINICAL TRIAL: NCT04999644
Title: Reduced Nicotine Cigarette Purchasing Decisions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00288837; R03DA054098-01 (NIH)
Record Dates: First submitted 2021-07-15; First posted 2021-08-11 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Full Nicotine Expectancy, Reduced Nicotine Dose (Experimental): Receive reduced nicotine cigarette expecting full
  Interventions: Drug: Reduced Nicotine Cigarettes; Behavioral: Average Nicotine Expectancy
- Full Nicotine Expectancy, Full Nicotine Dose (Experimental): Receive full nicotine cigarette expecting full
  Interventions: Drug: Full Nicotine Cigarettes; Behavioral: Average Nicotine Expectancy
- Reduced Nicotine Expectancy, Full Nicotine Dose (Experimental): Receive full nicotine cigarette expecting reduced
  Interventions: Drug: Full Nicotine Cigarettes; Behavioral: Very Low Nicotine Expectancy
- Reduced Nicotine Expectancy, Reduced Nicotine Dose (Experimental): Receive reduced nicotine cigarette expecting reduced
  Interventions: Drug: Reduced Nicotine Cigarettes; Behavioral: Very Low Nicotine Expectancy

INTERVENTIONS:
Drug: Full Nicotine Cigarettes — A full nicotine tobacco cigarette that will be smoked by participants
  Arms: Full Nicotine Expectancy, Full Nicotine Dose; Reduced Nicotine Expectancy, Full Nicotine Dose
Drug: Reduced Nicotine Cigarettes — A reduced nicotine tobacco cigarette that will be smoked by participants
  Arms: Full Nicotine Expectancy, Reduced Nicotine Dose; Reduced Nicotine Expectancy, Reduced Nicotine Dose
Behavioral: Average Nicotine Expectancy — Participant instructed the cigarette is "the same level of nicotine as your usual brand."
  Arms: Full Nicotine Expectancy, Full Nicotine Dose; Full Nicotine Expectancy, Reduced Nicotine Dose
Behavioral: Very Low Nicotine Expectancy — Participant instructed the cigarette is "a very low level of nicotine compared to your usual brand."
  Arms: Reduced Nicotine Expectancy, Full Nicotine Dose; Reduced Nicotine Expectancy, Reduced Nicotine Dose

SUMMARY:
The goal of this project is to experimentally evaluate how expectations about reduced-nicotine cigarettes as well as actual nicotine content interact to determine behavioral and subjective response for these novel products.

ELIGIBILITY:
Inclusion criteria:

* 21 years or older
* Smoke five or more cigarettes per day for the past six months
* Biological confirmation of cigarette use: have an expired carbon monoxide (CO) level of more than 8 ppm and a urinary cotinine level of more than 100 ng per milliliter at screening

Exclusion criteria:

* Intention to quit smoking in the next 30 days
* Weekly use of nicotine-containing products other than machine-manufactured combustible cigarettes
* Serious medical or psychiatric disorder precluding participation by study physician guidance
* Positive urine screening for illicit drugs other than cannabis or current substance use disorder
* Women who are pregnant, plan to become pregnant, or are breast-feeding
* Medical contraindications to receiving tobacco products

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Johnson, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Included in Analysis: This study used a within subjects design (i.e., all subjects were to receive all conditions, full and reduced nicotine tobacco cigarette). Twenty-one subjects completed the study.
Period: Overall Study
Arm/Group | Subjects Included in Analysis
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects Included in Analysis: This study used a within subjects design (i.e., all subjects were to receive all conditions). Twenty-one subjects completed the study.
Arm/Group | Subjects Included in Analysis
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Demand Intensity
Description: Consumption of cigarettes at unconstrained price as measured by an incentivized demand task. Minimum value is 0, maximum value is not constrained. Higher scores indicate more cigarette consumption at unconstrained price (a worse outcome).
Time Frame: Four times over approximately two weeks
Measure: Mean (Standard Error); unit: cigarettes
Arm/Group | Subjects Included in Analysis
Number analyzed (Participants) | 21
cigarettes
  Condition A: Told Full, Received Reduced | 6.48 (4.55)
  Condition B: Told Full, Received Full | 8.10 (6.61)
  Condition C: Told Reduced, Received Full | 7.81 (5.63)
  Condition D: Told Reduced, Received Reduced | 6.48 (4.91)

2. Primary Outcome: Demand Elasticity
Description: Changes in cigarette consumption with changes in price as measured by an incentivized demand task. There is no minimum or maximum value. Higher scores indicate greater cigarette price sensitivity (a better outcome). Values are log-transformed. Data are presented for all subjects with non-zero data (zero data cannot be analyzed with a demand function so elasticity cannot be generated)
Time Frame: Four times over approximately two weeks
Population: Data are presented for all subjects with non-zero data
Measure: Mean (Standard Deviation); unit: log(cigarettes/dollar)
Arm/Group | Subjects Included in Analysis
Number analyzed (Participants) | 21
log(cigarettes/dollar)
  Condition A: Told Full, Received Reduced: number analyzed (Participants) | 20
  Condition A: Told Full, Received Reduced | -1.31 (1.08)
  Condition B: Told Full, Received Full: number analyzed (Participants) | 20
  Condition B: Told Full, Received Full | -1.45 (0.50)
  Condition C: Told Reduced, Received Full: number analyzed (Participants) | 19
  Condition C: Told Reduced, Received Full | -1.57 (0.60)
  Condition D: Told Reduced, Received Reduced: number analyzed (Participants) | 18
  Condition D: Told Reduced, Received Reduced | -1.26 (1.17)

3. Secondary Outcome: Minnesota Nicotine Withdrawal Scale
Description: A subjective effect measure of nicotine withdrawal. Minimum value is 0, maximum value is 68. Higher scores indicate greater nicotine withdrawal (a worse outcome).
Time Frame: Post-cigarette administration four times over approximately two weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Included in Analysis
Number analyzed (Participants) | 21
units on a scale
  Condition A: Told Full, Received Reduced | 5.67 (6.95)
  Condition B: Told Full, Received Full | 5.14 (6.54)
  Condition C: Told Reduced, Received Full | 4.33 (4.95)
  Condition D: Told Reduced, Received Reduced | 6.24 (6.47)

ADVERSE EVENTS:
Time Frame: Approximately two weeks
Arm/Group | Subjects Included in Analysis
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04999644/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04999644/ICF_001.pdf